CLINICAL TRIAL: NCT00859833
Title: Effects of Body Mass Index on the Hyperemic Response to Regadenoson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sheldon Litwin, M.D., Professor of Medicine, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 31431
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Obesity; Endothelial Dysfunction; Decreased Vascular Flow
Keywords: adenosine; regadenoson; adenosine receptor subtypes
MeSH Terms: conditions — Obesity | interventions — Adenosine; regadenoson

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- myocardial perfusion reserve (Experimental): Myocardial perfusion reserve will be measured by quantifying myocardial blood flow using MRI at rest and then with each of 2 coronary vasodilators. Measurements are performed with first pass gadolinium perfusion (i.v. bolus injection of 0.02 or 0.03 mmol/kg of gadolinium). Each of the 2 drugs is given sequentially (30 minutes apart) in the same sequence in every patient. The shorter acting drug (adenosine) is given first so it has time to wear off before giving the second drug. It is ideal to measure MPR with each drug during the same imaging session so that there are no other clinical variables that change between the administration of the 2 agents. See below.
  Interventions: Drug: Adenosine; Drug: Regadenoson

INTERVENTIONS:
Drug: Adenosine — Myocardial perfusion reserve measured with quantitative MRI during adenosine infusion (0.14 mg/kg/min x 6 minutes).
  Other Names: adenoscan
Drug: Regadenoson — Myocardial perfusion reserve measured during regadenoson (0.4 mg/5 ml) bolus administration using quantitative perfusion MRI.
  Other Names: Lexiscan

SUMMARY:
We will test the hypothesis that a single dose of Regadenoson will produce equivalent degrees of coronary hyperemia in patients of widely different body size. This will be a prospective, open-label, comparative trial using MRI to measure myocardial perfusion reserve (ratio of myocardial blood flow with vasodilator to myocardial blood flow at rest) during sequential administration of the coronary vasodilators adenosine and regadenoson. Non-invasive MRI measurements of resting myocardial blood flow, and sequential measurements of blood flow during adenosine infusion (weight adjusted dosing) and then blood flow during regadenoson infusion (single, fixed dose. Blood flow measurements will be obtained sequentially and in the same sequence in each subject during a two hour MRI exam. 32 subjects will be recruited for this study. The first 2 will be for testing of the protocol. Inclusion criteria: 2 subjects for initial protocol evaluation, then 30 subjects with body mass index (BMI) between 18 and 40. Exclusions are pregnancy, renal dysfunction and claustrophobia.

DETAILED DESCRIPTION:
Introduction: Regadenoson (Lexiscan) is currently recommended for use as a targeted vasodilator in myocardial perfusion studies and is available as a single, fixed dose for all patients. Here we propose to compare the hyperemic response measured with MRI in subjects with a wide range of BMI 18-40.

MRI is an ideal test to compare the effects of regadenoson in patients with different body mass indices (BMIs). No radiation is used and multiple perfusion tests can be performed in close temporal sequence. Importantly, a number of researchers have shown the ability to obtain quantitative stress and rest myocardial blood flow values in the heart with MR imaging. This allows the calculation of myocardial perfusion reserve (MPR). Flow reserve measurements also can be done with dynamic PET, but not with SPECT. PET has the disadvantage of radiation exposure.

Regadenoson may be a more desirable agent for use with MRI than is adenosine. Adenosine requires the use of 2 intravenous lines, and the use of either a specialized, expensive, MRI-compatible infusion pump to deliver the drug, or long lengths of tubing to run to a pump outside the scanner room. Neither solution is ideal. Regadenoson does not require any such pumps or the starting of a second i.v.. The work here would accomplish 2 goals: 1) to demonstrate the feasibility of performing quantitative MRI perfusion measurements with regadenoson, and 2) to test whether a single dose of regadenoson produces maximal coronary hyperemia across a wide range of body sizes.

Study Design: This will be a prospective, open-label, study. The design is single group, one arm, 2 interventions in which we will compare MPR measured sequentially during adenosine and regadenoson using MRI. Non-invasive MRI measurements of resting flow, flow at adenosine stress, and flow at regadenoson stress will be obtained sequentially in each subject during a single two hour MRI exam. Each drug will be given in the same order to all subjects.

32 subjects will be recruited for this study. The first two subjects will be imaged only with resting perfusion, in order to determine optimal acquisition parameters for the study, and will not be used in the analysis. The main outcome measure is MPR with each agent.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-40 kg/m^2
* age 18-88

Exclusion Criteria:

* critically ill patients, patients on ventilators, patients with hypotension, asthmatics, and other patients whose medical care or safety may be compromised from undergoing an MRI examination will be excluded.
* Patients with claustrophobia will also be excluded.
* Also, anyone with contraindications to MRI (pacemaker, ICD, metal implants), pregnant subjects, minors, and prisoners will be excluded from this study.
* If subjects are over 60 or have any suspicion of abnormal kidney function, a blood test to determine GFR will be performed prior to imaging.
* Subjects with GFR < 30 will be excluded from the study.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon E Litwin, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] DiBella EV, Fluckiger JU, Chen L, Kim TH, Pack NA, Matthews B, Adluru G, Priester T, Kuppahally S, Jiji R, McGann C, Litwin SE. The effect of obesity on regadenoson-induced myocardial hyperemia: a quantitative magnetic resonance imaging study. Int J Cardiovasc Imaging. 2012 Aug;28(6):1435-44. doi: 10.1007/s10554-011-9949-4. Epub 2011 Oct 4. PMID 21968545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinics and by advertising within the hospital.
Groups:
- Adenosine Followed by Regadenoson: Myocardial perfusion reserve measured during adenosine infusion (140 ug/kg/min x 6 minutes). 30 minutes later regadenoson was given (0.4 mg) given as in i.v. bolus.
Period: Overall Study
Arm/Group | Adenosine Followed by Regadenoson
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adenosine Followed by Regadenoson: Myocardial perfusion reserve measured during adenosine infusion (140 ug/kg/min x 6 minutes). 30 minutes later regadenoson 0.4 mg given intravenous bolus.
Arm/Group | Adenosine Followed by Regadenoson
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.5)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion Reserve Measured by Quantitative Perfusion MRI (Ratio of Myocardial Blood Flow During Stress Over Myocardial Blood Flow at Rest)
Description: The ratio of myocardial blood flow during stress (with each vasodilator) divided by the myocardial flood flow at rest = myocardial perfusion reserve (MPR)
Time Frame: 2 hours
Population: Analysis was per protocol. All patients with analyzable data were included. 2/30 patients had technical problems with the MRI data that made their data unable to be analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Adenosine: Myocardial perfusion reserve measured during adenosine infusion (140 ug/kg/min x 6 minutes).
- Regadenoson: Regadenoson 0.5 mg i.v. bolus.
Arm/Group | Adenosine | Regadenoson
Number analyzed (Participants) | 28 | 28
ratio | 2.25 (0.59) | 2.44 (0.91)
Statistical Analysis 1: Comparison: Adenosine; Null hypothesis is that myocardial perfusion reserve (MPR) is not different when measured with adenosine or regadenoson in patients across a broad range of body sizes; Test type: Non-Inferiority or Equivalence — Power calculation for equivalence: SD for adenosine = 0.59, SD for regadenoson = 0.92, true difference between groups = 0.19. With n=28, DOF = 46. Power for equivalence (with alpha = 0.05) = 0.98585; p = 0.3617, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.6041 to 0.2241], Standard Deviation 0.7

ADVERSE EVENTS:
Arm/Group | Adenosine Followed by Regadenoson
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Due to technical problems, data from two of the 30 subjects was not usable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less